CLINICAL TRIAL: NCT01768221
Title: Caregiver Outlook: An Evidence-based Intervention for the Chaplain Toolkit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00039370
Record Dates: First submitted 2012-12-05; First posted 2013-01-15 (Estimated); Last update posted 2017-12-04 (Actual); Status verified 2017-08

CONDITIONS: Caregiver Wellbeing
Keywords: Palliative Care; Caregiver Outlook

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Caregiver intervention (Other)
  Interventions: Behavioral: Caregiver Intervention

INTERVENTIONS:
Behavioral: Caregiver Intervention — Participants will speak with a chaplain for three brief, 45 minute to one hour, sessions.
  The sessions will focus on topics of relationship life review, unresolved conflicts and issues of forgiveness, and future goals, lessons learned and legacy.
  In the week following the third session, the chaplain will call participants for a brief check in. This call will include no new intervention content, rather it provides an opportunity for participants to mention any additional thoughts or concerns they want to discuss with the chaplain interventionist.

SUMMARY:
This one-arm pilot study will evaluate the feasibility and acceptability of Caregiver Outlook, a manualized chaplain-led intervention to improve the well-being of caregivers of seriously ill patients.

Study Activities and Population Group:

The investigators anticipate enrolling 36 informal caregivers (adults) through DUMC providers and/or self-referral. Potential subjects will be screened for study eligibility, consented if eligible and interested, and one week later administered a baseline survey by phone. Next, the chaplain-led intervention will be delivered by phone in three one-hour sessions, spanning a one month window. After session 3, subjects will receive a check-in phone call to briefly discuss their any additional thoughts, questions or concerns they may have. Sessions will be audio recorded. After intervention completion, follow-up surveys will be administered by phone at two points in time.

Data Analysis and Risk/Safety Issues:

This is a mixed-methods study involving qualitative thematic analysis and survey data, collected from the adult caregiver subjects. There are no known physical risks to participation, and the study team will work to ensure confidentiality and data safety/integrity.

DETAILED DESCRIPTION:
Tasks of preparation and completion - reviewing one's life, assessing unfinished business, addressing relationship conflicts, offering or receiving forgiveness, and identifying wisdom gained and future goals - are associated with quality in both palliative care and chaplaincy care. The consequences are dramatic when preparation and completion at the very end of life are not achieved, and unmet needs in these domains influence caregiver experience earlier and throughout longer periods during the trajectory of serious illness.

Efforts to improve the caregiver experience have tended to focus on skill-building and self-efficacy for providing care, including patient pain and symptom management, and caregiver coping. However, less is known about effective ways to address other elements of caregivers' experience that may influence well-being and capacity to care, namely the meaning caregivers' ascribe to their caregiving role. Research shows caregivers with higher sense of meaning report lower subjective caregiver burden. In palliative care, the important tasks of caregiver preparation and completion are tools through which caregivers engage in meaning-making, identifying purpose, and connecting with what is held sacred.

These tasks are central to patient and family definitions of quality at end-of-life, and the goals and skills of healthcare chaplaincy. Addressing issues of meaning, exploring relational well-being, and supporting caregiver's own sense of loss and hope is at the heart of chaplaincy care. Professional chaplaincy uses narrative pastoral care to help patents, families, significant others, and staff focus on meaning-making and quality of life in the midst of health celebrations, changes, crises, and loss. Clinical chaplains focus on caregiver's specific concerns, values, beliefs, and practices that enhance caring with integrity and authenticity for the purpose of ongoing spiritual assessment and pastoral care planning.

However, both the manner and extent to which caregiver concerns are addressed vary based on family and patient circumstance, time available, and individual chaplain skill. The majority of chaplain's approaches to these concerns have not been delivered or evaluated in a manualized format. The chaplaincy profession's evidence base would be strengthened by systematically exploring the content of such an approach, its impact on caregiver health outcomes, and the ways a manualized intervention approach ("Caregiver Outlook") may serve as a foundation for the chaplain's future teaching, practicing, and researching of systematized spiritual assessment and care planning processes.

The investigators propose a one-arm pilot trial to evaluate the feasibility and acceptability of a chaplain-led preparation and completion intervention, and also to examine effect sizes on health outcomes. Results will permit feasibility and acceptability evaluation of an evidence-based tool for addressing and assessing caregivers' spiritual strengths and experiences of suffering in palliative care. The project will serve as a foundation to understand integration of the central tasks of preparation and completion with other approaches to spiritual assessment and pastoral care planning. Finally, results will provide preliminary data for future large-scale randomized control trials of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older;
* Able to read and speak English, as assessed by study staff;
* Has a phone (or has access to a phone);
* Provides daily care to a spouse, parent, or child with advanced disease - "care" includes day-to-day assistance and support, and "advanced disease" will be confirmed by a healthcare provider OR by a Palliative Performance Scale (PPS) score below 70%, as assessed by the caregiver (the patient will not be assessed);
* Cognitively capable to give informed consent, as determined by staff.

Exclusion Criteria:

* Caregivers of patients in hospice at time of consent (but if a patient enters hospice during the study, the caregiver may continue).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Feasibility and acceptability of a chaplain-led intervention | 8 weeks
  Assess caregivers' spiritual strengths and experiences by conducting surveys and interviews to measure change in anxiety, preparation and completion, grief, depression and caregiver reactions at baseline and post intervention at 6 weeks, and 8 weeks.

SECONDARY OUTCOMES:
Caregiver Outlook intervention qualitative discussion theme content and variation | Baseline (week 1)
  The study will examine Caregiver Outlook intervention qualitative discussion theme content and variation associated with gender, ethnicity, SES, type and stage of illness, and spirituality measures.
Intervention responses | Weeks 2-5
  The study will examine intervention responses for themes that lead to integration with spiritual assessment and other approaches to chaplaincy care and pastoral care planning.
Evaluate and establish effect sizes associated with Caregiver Outlook on caregiver anxiety, depression, anticipatory grief, quality of life, and burden. | Baseline (week 1), Followup (Week 6), Followup 2 (Week 8)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Steinhauser, PhD, Principal Investigator — General Internal Medicine/Durham VA
Locations (1):
- Duke University Health System, Durham, North Carolina, United States